CLINICAL TRIAL: NCT00367692
Title: An Exploratory, Double Blind, Placebo-controlled, Randomized, Single-dose, Cross-over, Proof of Mechanism Study of Orally Administered PSI-697 in Patients With Scleritis
Brief Title: Study Evaluating PSI-697 in Patients With Scleritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 3165A1-106
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Scleritis
Keywords: Scleritis
MeSH Terms: conditions — Scleritis | interventions — 2-(4-chlorobenzyl)-3-hydroxy-7,8,9,10-tetrahydrobenzo(H)quinoline-4-carboxylic acid

INTERVENTIONS:
Drug: PSI-697

SUMMARY:
To evaluate the safety of an orally administered single dose of PSI-697 in subjects with scleritis, as a model of inflammatory disease. To evaluate by in vivo confocal microscopy (IVCM) the effect of a single dose of PSI-697 on leukocyte rolling in the scleral blood vessels of subjects with scleritis.

ELIGIBILITY:
Inclusion: Age 18 or higher; A negative urine pregnancy test at screening for female subjects; Female subjects must be postmenopausal or surgically sterile.

Exclusion: Isolated episcleritis; Isolated posterior scleritis; Infectious scleritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-09; Study Completion 2007-04

PRIMARY OUTCOMES:
To evaluate by IVCM the effect of a single dose of PSI-697 on leukocyte rolling in scleral blood vessels of subjects with scleritis.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer